CLINICAL TRIAL: NCT01692691
Title: Phase II Trial of Sequenced Chemotherapy With Dacarbazine and Carmustine With Neulasta® Support in Previously Treated Metastatic Melanoma
Brief Title: Dacarbazine and Carmustine in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decision
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-10
Record Dates: First submitted 2012-08-29; First posted 2012-09-25 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Melanoma Metastatic
Keywords: Melanoma Metastatic
MeSH Terms: interventions — Dacarbazine; Carmustine; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacarbazine, carmustine, neulasta (Experimental): Dacarbazine IV - Day 1; Carmustine IV - Day 2; Neulasta SC - Day 3
  Interventions: Drug: Dacarbazine; Drug: Carmustine; Drug: Neulasta

INTERVENTIONS:
Drug: Dacarbazine — Dacarbazine IV - Day 1
  Other Names: DTIC
Drug: Carmustine — Carmustine IV- Day 2
  Other Names: BCNU
Drug: Neulasta — Neulasta SC - Day 3
  Other Names: pegfilgrastim

SUMMARY:
The purpose of this study is to determine whether dacarbazine and carmustine at the doses and schedule used in this study will help to increase tumor shrinkage.

DETAILED DESCRIPTION:
In this phase II trial, patients with stage IV melanoma will be treated with dacarbazine and carmustine commonly used in this cancer, but given using a schedule that might theoretically improve on this combination. Patients on this study will be assessed in terms of toxicity, response rate, median duration of response, median time to disease progression, and median survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically-proven diagnosis of metastatic malignant melanoma which has progressed on at least one prior systemic therapy.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 and estimated survival of at least 3 months.
3. Patients must be felt to have recovered from effects of prior cancer therapy, such as past expected leukocyte nadir for chemotherapy (> 2 weeks).
4. Absolute granulocyte count of at least 1500/mm3; hemoglobin of at least 9 gm/dl; platelet count of at least 100,000/mm3; bilirubin must be less than 1.5 mg/dl; ALT and AST must be less than 3 times the upper limit of normal; creatinine must be less than or equal to 1.8 mg/dl.
5. Women of childbearing potential must have a negative pregnancy test and adequate precautions to prevent pregnancy during treatment must be taken.
6. Patient consent must be obtained prior to entrance onto study.
7. Patients must have no evidence of significant cardiovascular disease including history of recent (< 6 months) myocardial infarction, uncompensated congestive heart failure, uncontrolled angina or cerebrovascular accident.

Exclusion Criteria:

1. Evidence of significant cardiovascular disease including history of recent (< 6 months) myocardial infarction, uncompensated congestive heart failure, uncontrolled angina, or cerebrovascular accident.
2. Prior history of psychiatric disorder that could be exacerbated by or which could preclude completion of this therapy.
3. Pregnancy or lactation.
4. Prior chemotherapy with carmustine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, FNP, Study Director — CTCA
Locations (1):
- Western Regional Medical Center, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dacarbazine Carmustine: All patients received chemotherapy with Dacarbazine and Carmustine
Period: Overall Study
Arm/Group | Dacarbazine Carmustine
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Received Treatment: Dacarbazine Carmustine participants
Arm/Group | Received Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival of patients with Stage IV melanoma who have had disease progression on at least one prior systemic therapy
Time Frame: 8 weeks
Population: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Groups:
- Participants 8 Week Survival.: Number of participants who received Dacarbazine + Carmustine Progression Free survival at 8 weeks
Arm/Group | Participants 8 Week Survival.
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate
Description: To determine the response rate after being treated with Dacarbazine Carmustine
Time Frame: 8 weeks
Population: as for outcome 1
Groups:
- Response Rate: Dacarbazine Carmustine
Arm/Group | Response Rate
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Duration of Response
Description: To determine the median duration of response for patients who received Dacarbazine and Carmustine
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Dacarbazine Carmustine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Received Treatment: Number of Participants who received Dacarbazine Carmustine
Arm/Group | Received Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Received Treatment (N=1)
Nausea (Gastrointestinal disorders) | 0
Arthalgia (General disorders) | 0
gastroesophageal reflux (Gastrointestinal disorders) | 0
Leukopenia (Investigations) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes